CLINICAL TRIAL: NCT03501004
Title: The Study of Acupuncture on Vascular and Functional Neuroimaging in Parkinson's Disease Patients With Sleep Disorders
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tsinghua University (Other)
Responsible Party: Principal Investigator, Yu Ma, Associate Professor, Tsinghua University
Allocation: Randomized | Model: Single Group | Masking: Triple | Purpose: Treatment
Other Study IDs: QHDXYQYY20180001
Record Dates: First submitted 2018-03-25; First posted 2018-04-18 (Actual); Last update posted 2021-04-12 (Actual); Status verified 2021-04

CONDITIONS: Acupuncture; Parkinson's Disease; Sleep Disorders; Neuroimaging
MeSH Terms: conditions — Parkinson Disease; Sleep Wake Disorders

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- The Acupuncture Group (Experimental): Sterile acupuncture needles for single use will be used.The intervention is going to be executed using the acupuncture points GV14（Dazhui）and GB20 (Fengchi) for 20 minutes.The acupuncture needles will be inserted to a depth of 0.8 to 1 cm using GV14（Dazhui）and GB20 (Fengchi).
  Interventions: Device: Sterile acupuncture needles for single use
- The Sham Acupuncture Group (Sham Comparator): Sterile acupuncture needles for single use will be used.The sham acupuncture group's acupuncture needles will be inserted to a depth of 0.1 to 0.2 cm with nonacupuncture points located 0.5 cm in lateral to the real acupoint or to the right for midline points for 20 minutes.
  Interventions: Device: Sterile acupuncture needles for single use

INTERVENTIONS:
Device: Sterile acupuncture needles for single use — Sterile acupuncture needles for single use are made by China Beijing Zhongyan Taihe Medical Instrument Limited Company.Acupuncture needles' specifications are 0.25mm*25mm.

SUMMARY:
The purpose of the study is to compare vascular and functional neurological changes of acupuncture in patients with Parkinson's Disease and Sleep Disorders. In the randomized controlled clinical trial study, patients meeting the criteria for inclusion will be randomly enrolled and divided into two groups in a 1:1 ratio: the acupuncture group and the sham acupuncture group. The intervention is going to be executed using the acupoints GV14（Dazhui）and GB20 (Fengchi).The acupuncture needles will be inserted to a depth of 0.8 to 1 cm using GV14（Dazhui）and GB20 (Fengchi) in the acupuncture group. The sham acupuncture group's needles will be inserted to a depth of 0.1 to 0.2 cm with nonacupuncture points located 0.5 cm in lateral to the real acupoint or to the right for midline points.During the study, researchers will observe changes in cerebral blood vessels and neuroimaging before and after acupuncture in the two groups. Using multimodal fusion advanced vascular-neuronal imaging techniques could evaluate the effect of acupuncture on brain blood vessels and function in patients with Parkinson's disease and Sleep Disorders and provide an objective neuroimaging basis for assessing the effectiveness of acupuncture.

DETAILED DESCRIPTION:
Neuroimaging assessment:Subjects are keeping awake, resting flat on the examination table, using rubber earplugs to reduce noise, using foam headbands to fix head movement artifacts, closing eyes to calm breathing, fixing the head and minimizing head and other parts of the initiative and passive exercise.At the same time, it is required not to carry out any thinking activities. After the subject is familiar with the environment, it begins to scan and conduct a comprehensive MRI scan before and after the acupuncture needling.

ELIGIBILITY:
Inclusion Criteria:

1. meeting the above diagnostic criteria for Parkinson's disease and Sleep Disorders;
2. Hoehn-Yahr grade 2-3;
3. Those who voluntarily participate in the project while he/she or his/her guardian sign an informed consent form;
4. Those who have had a junior high school education or above and have a correct understanding of clinical acupuncture research significance.

Exclusion Criteria:

1. Accompanied with sleep apnea syndrome, sleep-behavioral disorders such as sleep-breathing disorders, and other system diseases that cause sleep disorders, such as anemia and other hematological diseases, hypothyroidism, severe heart and lung diseases, tumors, liver and kidney diseases;
2. History of drug use or alcohol addiction, psychosis and sedation for painful illnesses;
3. Severe cognitive impairments and failure to complete scale assessments;
4. There are barriers to communication and communication that affect the evaluation of research, such as speech, vision, hearing and other serious damage to patients;
5. Allergic to needles or alcohol;
6. Those who cannot perform MRI scans, such as claustrophobia.

Ages: 40 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2018-06-01 (Actual); Primary Completion 2020-06-30 (Actual); Study Completion 2020-09-30 (Actual)

PRIMARY OUTCOMES:
Cerebral blood flow data change | Through once acupuncture completion, 30 minutes
  Neuroimaging assessment by 3D SNAP-MRA

SECONDARY OUTCOMES:
Parkinson's Disease Sleep Scale | Through once acupuncture completion, 30 minutes
  Scale evaluation.Scale Range:0-150.Higher values represent a better outcome.
Pittsburgh Sleep Quality Index | Through once acupuncture completion, 30 minutes
  Scale evaluation.Scale Range:0-21.Higher values represent a worse outcome.
Epworth Sleepiness Scale | Through once acupuncture completion, 30 minutes
  Scale evaluation.Scale Range:0-24.Higher values represent a worse outcome.
Unified Parkinson's Disease Rating Scale | Through once acupuncture completion, 30 minutes
  Scale evaluation.Scale Range:0-149.Higher values represent a worse outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Yuqi Zhang, Study Chair — Tsinghua University Yuquan Hospital
Locations (1):
- Tsinghua University Yuquan Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data for all primary and secondary outcome measures will be made available.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Data will be available within 12 months of study completion.
Access Criteria: Data access requests will be reviewed by an external Independent Review Panel. Requestors will be required to sign a Data Access Agreement.